CLINICAL TRIAL: NCT00949052
Title: Radiation Sensitivity, DNA Repair, and Second Cancers.
Brief Title: Genetic Susceptibility and Risk of Second Cancers in Patients Who Have Undergone Stem Cell Transplant for Cancer
Status: Terminated | Type: Observational
Why Stopped: Low accrual
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Debra Friedman, Associate Professor of Pediatrics, Vanderbilt University Medical Center
Other Study IDs: VICC REACH 0901; P30CA068485 (NIH); FHCRC-2023 (Other: Fred Hutchinson Cancer Research Center); IRB# 090032 (Other: Vanderbilt University)
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Cancer
Keywords: cancer survivor; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Hodgkin lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; recurrent/refractory childhood Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); atypical chronic myeloid leukemia, BCR-ABL negative; blastic phase chronic myelogenous leukemia; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood chronic myelogenous leukemia; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; juvenile myelomonocytic leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; childhood myelodysplastic syndromes; chronic eosinophilic leukemia; primary myelofibrosis; chronic neutrophilic leukemia; de novo myelodysplastic syndromes; disseminated neuroblastoma; myelodysplastic/myeloproliferative neoplasm, unclassifiable; poor prognosis metastatic gestational trophoblastic tumor; previously treated childhood rhabdomyosarcoma; previously treated myelodysplastic syndromes; recurrent Wilms tumor and other childhood kidney tumors; recurrent childhood rhabdomyosarcoma; recurrent neuroblastoma; recurrent ovarian epithelial cancer; recurrent ovarian germ cell tumor; recurrent malignant testicular germ cell tumor; secondary myelodysplastic syndromes; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; stage III malignant testicular germ cell tumor; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; refractory multiple myeloma
MeSH Terms: conditions — Neoplasms; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Recurrence; Mycosis Fungoides; Sezary Syndrome; Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelomonocytic, Juvenile; Leukemia, Myeloid, Acute; Leukemia, Hairy Cell; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Neutrophilic, Chronic; Myeloproliferative Disorders; Wilms Tumor; Neuroblastoma; Carcinoma, Ovarian Epithelial; Testicular Neoplasms; Multiple Myeloma; Breast Neoplasms | interventions — Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA analysis
Genetic: polymorphism analysis
Other: laboratory biomarker analysis
Other: medical chart review
Other: questionnaire administration
Procedure: assessment of therapy complications
Procedure: evaluation of cancer risk factors

SUMMARY:
RATIONALE: Identifying genes that increase a person's susceptibility to second cancers may help the study of cancer treatment.

PURPOSE: This study is looking at genetic susceptibility and risk of second cancers in patients who have undergone stem cell transplant for cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether genetic susceptibility (e.g., inherited differences in radiation sensitivity to normal tissue or genes of xenobiotic metabolism, nucleotide provision, or DNA repair) to the carcinogenic effects of radiotherapy, tobacco, and UV light modifies the risk of second malignant neoplasms (SMN) in patients with cancer treated with hematopoietic stem cell transplantation (HSCT).

Secondary

* Measure inherent sensitivity to radiotherapy via G_2 chromosome radiation sensitivity assay using B-cell lymphoblastoid cell lines derived from pre-HSCT cryopreserved peripheral blood mononuclear cells of patients with and without SMN.
* Measure the frequency of allelic variants of genes involved in xenobiotics metabolism, DNA repair, and provision of nucleotide pool and compare the frequencies among patients with and without SMN, determine the transmission of specific alleles of these genes from parents to patients, and correlate allelic variants of DNA repair and nucleotide provision in genes with in vitro radiation sensitivity.
* Evaluate the role of potentially carcinogenic environmental exposures (tobacco and sun light) pre- or post-HSCT in the risk of SMN and examine the association of these exposures with SMN and the interaction of these exposures with allelic variants of genes involved in xenobiotic metabolism, nucleotide provision, and DNA repair.

OUTLINE: Patients complete self-reported questionnaires and medical records are reviewed to collect information on UV light and tobacco exposure pre- and post-transplantation. Information is analyzed for association with second malignancy neoplasms.

Blood samples are collected from patients pre-hematopoietic stem cell transplantation and from their parents (when available) or other first-degree relatives for genetic biomarkers of susceptibility to second malignancies, DNA repair and provision nucleotide, genetic susceptibility to toxicity from combined cancer therapies, and environmental carcinogens.

PROJECTED ACCRUAL: A total of 1,000 patients (800 patients without second malignant neoplasms [SMN] and 200 patients with SMN) will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

CASES are those who:

* Survived at least 100 days post-hematopoietic stem cell transplantation (HSCT).
* Developed an SMN after that time point.
* And received TBI as part of the preparative regimen.

CONTROLS are randomly selected:

* In a 4:1 ratio to cases from the same cohort of 100 day + survivors of HSCT who received TBI.
* Controls will be matched to the cases by race and primary diagnosis.
* In addition, they must have survived for at least the elapsed time between the case's HSCT and the secondary cancer, without development of an SMN.
* We are matching on primary diagnosis, as genotype or radiation sensitivity may predispose to specific primary cancers, as well as the SMNs.
* We are matching on race, as allele frequencies vary widely across ethnic groups.

Exclusion Criteria:

* Did not survive at least 100 days post-hematopoietic stem cell transplantation (HSCT).
* Did not develop an SMN after that time point.
* Did not receive TBI as part of the preparative regimen.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who survived 100 days post-hematopoietic stem cell transplantation (HSCT)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Genetic susceptibility to the carcinogenic effects of radiotherapy, tobacco, and UV light and risk of second malignant neoplasms (SMN) | At study entry

SECONDARY OUTCOMES:
Radiation sensitivity in B-cell lymphoblastoid cells | At study entry
Allelic variants of genes involved in xenobiotics metabolism, DNA repair, and provision of nucleotide pool of patients with SMN compared to their first-degree relatives and patients without SMN | At study entry
Role of potentially carcinogenic environmental exposures (tobacco and sun light) pre- and post-HSCT in the risk of SMN | At study entry

CONTACTS AND LOCATIONS:
Overall Officials: Debra L. Friedman, MD, MS, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States